CLINICAL TRIAL: NCT00798252
Title: A Phase I, Multi-arm, Dose Escalation Study of Brivanib Alaninate Combined With Several Chemotherapy Regimens in Subjects With Solid Tumors
Brief Title: Ascending Multiple-Dose Study of Brivanib Alaninate in Combination With Chemotherapeutic Agents in Subjects With Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA182-030; 2007-005097-31 (EudraCT Number)
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Advanced Cancer
Keywords: metastatic, chemotherapy combination
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Capecitabine; Doxorubicin; ixabepilone; Docetaxel; Paclitaxel; brivanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm A (Capecitabine + Brivanib alaninate) (Experimental)
  Interventions: Drug: Capecitabine; Drug: Brivanib alaninate
- Arm B (Doxorubicin + Brivanib alaninate) (Experimental)
  Interventions: Drug: Doxorubicin; Drug: Brivanib alaninate
- Arm C (Ixabepilone + Brivanib alaninate) (Experimental)
  Interventions: Drug: Ixabepilone; Drug: Brivanib alaninate
- Arm D (Docetaxel + Brivanib alaninate) (Experimental)
  Interventions: Drug: Docetaxel; Drug: Brivanib alaninate
- Arm E (Paclitaxel + Brivanib alaninate) (Experimental)
  Interventions: Drug: Paclitaxel; Drug: Brivanib alaninate

INTERVENTIONS:
Drug: Capecitabine — Tablets, Oral, Dose escalation to a MTD from a starting dose of 850 mg/m², twice a day (BID) x 14d per cycle, until disease progression
  Other Names: Xleoda®
  Arms: Arm A (Capecitabine + Brivanib alaninate)
Drug: Doxorubicin — IV, Dose escalation to a MTD from a starting dose of 40 mg/m², Q3wks, until disease progression
  Other Names: Adriamycin®
  Arms: Arm B (Doxorubicin + Brivanib alaninate)
Drug: Ixabepilone — IV, Dose Escalation to a MTD from a starting dose of 32 mg/m², Q3wks, until disease progression
  Other Names: IXEMPRA®; BMS-247550
  Arms: Arm C (Ixabepilone + Brivanib alaninate)
Drug: Docetaxel — IV, Dose escalation to an MTD from a starting dose of 60 mg/m², Q3wks, Until disease progression
  Other Names: Taxotere®
  Arms: Arm D (Docetaxel + Brivanib alaninate)
Drug: Paclitaxel — IV, Dose escalation to an MTD from a starting dose of Paclitaxel 135 mg/m², Q3wks, Until disease progression
  Other Names: Taxol®
  Arms: Arm E (Paclitaxel + Brivanib alaninate)
Drug: Brivanib alaninate — Tablets, Oral, Dose escalation to a MTD from a starting dose of 400 mg, daily (QD), until disease progression
  Other Names: BMS-540215

SUMMARY:
To determine safety and maximum tolerated dose of brivanib alaninate when administered in combination with capecitabine, doxorubicin, ixabepilone, docetaxel and paclitaxel chemotherapy to subjects with advanced or metastatic solid tumors

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Histologic/cytologic diagnosis of advanced or metastatic solid tumors
* Life expectancy >= 3 months
* Able to swallow tablets/capsules

Exclusion Criteria:

* Pregnant or breastfeeding women
* No more than 4 previous chemotherapy regimens in the advanced or metastatic setting (excluding prior adjuvant or hormonal / immuno / biologic antibody therapies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2009-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
To determine safety and the maximum tolerated dose of brivanib alaninate when administered in combination with capecitabine, doxorubicin, ixabepilone, docetaxel and paclitaxel chemotherapy to subjects with advanced or metastatic solid tumors | Every 21 days until the maximum tolerated dose (MTD) for each combination of brivanib is reached

SECONDARY OUTCOMES:
To describe the anti-tumor activity of brivanib alaninate combination with the different chemotherapeutic regimens: capecitabine, doxorubicin, ixabepilone, docetaxel, and paclitaxel | Every 21 days
To assess the effect each of capecitabine, doxorubicin, ixabepilone, docetaxel, and paclitaxel on the pharmacokinetics of BMS-540215 (active moiety of brivanib pro-drug) at the MTD | Cycle 1D21, Days 1, 2, 3, 8 of Cycles 1 & 2
To assess the effect of brivanib alaninate on the pharmacokinetics each of capecitabine, doxorubicin, ixabepilone, docetaxel, and paclitaxel chemotherapy regimens at the MTD | Cycle 1D21, Days 1, 2, 3, 8 of Cycles 1 & 2

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (3):
  - Usc/Norris Comprehensive Cancer Center, Los Angeles, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
- Canada (2):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Toronto, Ontario

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx